CLINICAL TRIAL: NCT03563625
Title: The Effect of Local Wound Infiltration Versus Caudal Block on Wound Infection and Healing After Inguinal Herniotomy Paediatrics
Brief Title: Local Wound Infiltration Versus Caudal Block on Wound Infection and Healing in Paediatrics Inguinal Herniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050103846/11-4-2017
Record Dates: First submitted 2017-12-01; First posted 2018-06-20 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Healing Surgical Wounds
Keywords: Local anesthetic; Hernioraphy; Wound healing
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: The patients will be classified randomly into two groups using closed envelope technique, 25 patients each:
  Group L: 25 patients will receive 1mg/kg bupivacaine 0.25% (diluted as 1ml bupivacaine + 1ml normal saline) by local infiltration in the wound before closure of the skin and subcutaneous.
  Group C: 25 patients will receive caudal block with 1mg/kg bupivacaine 0.25%.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinded to procedure done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block (Active Comparator): Caudal block with 1mg/kg bupivacaine 0.25%.
  Interventions: Procedure: Caudal block; Drug: Bupivacaine
- Wound infiltration (Active Comparator): Local wound infiltration with 1mg/kg bupivacaine 0.25%.
  Interventions: Procedure: Wound infiltration; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Caudal block — Caudal block/bupivacaine 0.25%
  Arms: Caudal block
Procedure: Wound infiltration — Local anesthetic wound infiltration/bupivacaine 0.25%
  Arms: Wound infiltration
Drug: Bupivacaine — bupivacaine

SUMMARY:
The aim of the present study is to assess effect of local wound infiltration in comparison with caudal block by bupivacaine 0.25% after inguinal herniotomy in pediatrics on: Wound infection and healing (primary outcome) and postoperative analgesia (secondary outcome).

DETAILED DESCRIPTION:
THE EFFECT OF LOCAL WOUND INFILTERATION VERSUS CAUDAL BLOCK ON WOUND INFECTION AND HEALING AFTER INGUINAL HERNIOTOMY IN PAEDIATRICS

INTRODUCTION Since the introduction of cocaine in 1884, local anesthetics have been used as a mainstay of pain management. However, numerous studies over the past several decades have elucidated the supplemental role of local anesthetics as antimicrobial agents. In addition to their anesthetic properties, medications, such as: bupivacaine and lidocaine have been shown to exhibit bacteriostatic, bactericidal, fungistatic, and fungicidal properties against a wide spectrum of microorganisms.(1) Johnson et al.(2)made a comprehensive literature search using MEDLINE 1950-present for in vitro and in vivo studies pertaining to the antimicrobial activity of various local anaesthetics on a broad range of bacterial and fungal pathogens. Studies testing the effect on microbial growth inhibition of local anaesthetics alone and in combination with other agents, such as: preservatives and other medications, as well as the effect of conditions, such as: concentration and temperature were included for review. Evidence suggests that local anesthetics as a class possess inherent antimicrobial properties against a wide spectrum of human pathogens. Limited studies attribute the mechanism of action of antimicrobial activity of local anesthetics to a disruption of microbial cell membrane permeability, leading to leakage of cellular components and subsequent cell lysis.(2) Multiple local anesthetics at concentrations typically used in the clinical setting (e.g.:- bupivacaine 0.125%-0.75%; lidocaine 1%-3%) inhibit the growth of numerous bacteria and fungi under various conditions. Different local anesthetics showed various degrees of antimicrobial capacity; bupivacaine and lidocaine, for example, inhibit growth to a significantly greater extent than does ropivacaine.(2) In 1943 Lofgren (3) developed lidocaine. This was an amide and had a low risk of allergic reactions in comparison to ester local anesthetics. This was followed by mepivacaine (1957), prilocaine (1960), bupivacaine (1963), ropivacaine (1997) and levobupivacaine (2000).(3) Bupivacaine has been used in clinical practice for more than 40 years. It is remarkably stable in solution and is commercially available in 0.25% and 0.5% solutions (with and without epinephrine). Spinal heavy bupivacaine (0.5% bupivacaine + 6% glucose) is also manufactured. It is four times more potent than lidocaine. Therefore, 0.25% bupivacaine is equipotent with 1% lidocaine. Bupivacaine is particularly cardiotoxic and should never be used in Biers blocks. Bupivacaine binds tightly to tissues and thus has a long duration of action (up to 24 hours in some cases). Adding epinephrine will decrease its toxicity by delaying the drug absorption but, will have minimal effect on the duration of the block.(3)

The recommended maximum safe doses of bupivacaine are as follows:

BUPIVACAINE WITHOUT EPINEPHRINE ------- 2.0 mg/kg BUPIVACAINE WITH EPINEPHRINE ------- 2.5 mg/kg.(3) Caudal anesthesia is one of the most used-popular regional blocks in children. This technique is a useful adjunct during general anesthesia and for providing postoperative analgesia after infraumbilical operations. The quality and level of the caudal blockade is dependent on the dose, volume, and concentration of the injected drug.(4) Prophylactic analgesia with local anesthetics is an attractive concept, especially in pediatric practice, because the evaluation of pain can be very challenging in young children.(5) In contrast to opioids, local anesthetics can be administered safely, and in recent guidelines regional anaesthesia is accepted as the cornerstone of post-operative pain relief in the pediatric patients.(6) Although regional anaesthesia holds a good safety record overall, the global experience with pediatric regional anaesthesia is still quite low; even the most commonly performed procedure, caudal block, represents only 2.5% of all central neuroaxial blocks performed.(7,8) Determining the risk-benefit ratio is rather difficult for techniques that are relatively rarely performed. Wound infiltration can produce reliable analgesia for superficial skin surgery. Infiltration itself is extensively used by pediatricians, surgeons and emergency physicians for skin laceration repair or minor superficial surgery.(5) Several studies have compared the local anesthesia so far, including: ilio-inguinal and iliohypogastric nerve block plus subcutaneous injection by the surgeon against the caudal anesthesia.(9,10) But to our knowledge, there is still no study comparing the local wound infiltration by itself and caudal anesthesia for postoperative analgesia as regard their effect on wound infection and healing.

AIM OF THE WORK The aim of the present study is to assess effect of local wound infiltration in comparison with caudal block by bupivacaine 0.25% after inguinal herniotomy in pediatrics on: Wound infection and healing (primary outcome) and postoperative analgesia (secondary outcome).

PATIENTS After approval of ethical committee faculty of medicine, University of Alexandria, a prospective interventional concealed randomized clinical study which will include 50 children (calculated by department of community medicine) aged 2 months-1 year admitted to the Pediatrics Surgery Department of Alexandria University Hospitals for elective inguinal herniotomy surgery, and an informed written consent will be taken from the parents or the guardians.

All patients will be selected to be grade I or II according to American Society of Anesthesiologists (ASA) classification

The patients will be classified randomly into two groups using closed envelope technique, 25 patients each:

Group L: 25 patients will receive 1mg/kg bupivacaine 0.25% (diluted as 1ml bupivacaine + 1ml normal saline) by local infiltration in the wound before closure of the skin and subcutaneous.

Group C: 25 patients will receive caudal block with 1mg/kg bupivacaine 0.25%.

Exclusion criteria included:

* History of developmental delay or mental retardation.
* Diabetes mellitus type I.
* Known allergy or contraindication to any local anesthetics.
* Known congenital anomaly in the inguinal region.
* Any patient who will develop any infections postoperatively (respiratory infection, urinary infection) other than wound infection will be excluded.

METHODS

All patients will be subjected to the following:

A) Pre-operative visit:

Each patient will be visited the day before surgery for the following:

* Proper evaluation by history taking from parents, clinical examination and laboratory investigations.
* Explanation of the technique of postoperative analgesia to the parents and explain to them that the wound will be observed postoperatively for signs of inflammation and infection.

B) Pre-medication:

Paracetamol suppository 40mg/kg will be given half an hour before surgery.

C) Anaesthesia:

* All patients will be monitored for:

  * Heart rate (beats/minute) through continuous ECG tracing (lead II).
  * Non-invasive arterial blood pressure (mmHg).
  * Arterial oxygen saturation using pulse oximetry (%).
* Induction of general anaesthesia will be achieved with 8% sevoflurane in 100% oxygen.
* After securing an IV line with cannula, all patients will receive fentanyl 1mcg /kg.
* Laryngeal mask air way of proper size will be inserted under adequate depth of anaesthesia.
* Anaesthesia will be maintained with sevoflurane with concentration maintaining adequate depth of anaesthesia.
* At the end of procedure and before application of stitches, bupivacaine 0.25% will be infiltrated in the skin and subcutaneous layer in group L, and caudal block will be performed in group C; at the end of surgery inhalational anaesthetics will be stopped; laryngeal mask will be removed when patient is fully conscious.
* Postoperative pain will be assessed using the Faces Legs Activity Cry Consolability tool (FLACC, 0- 10) at 15 min, 1, and 3 h after operation.(11) Table (I): FLACC scale (Behavioral observation pain rating scale) Categories Scoring 0 1 2 Face No particular expression or smile; disinterested Occasional grimace or frown, withdrawn Frequent to constant frown, clenched jaw, quivering chin Legs No position or relaxed Uneasy, restless, tense Kicking, or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting back and forth, tense Arched, rigid, or jerking Cry No crying (awake or asleep) Moans or whimpers, occasional complaint Crying steadily, screams or sobs, frequent complaints Consolability Content, relaxed Reassured by occasional touching, hugging, or talking to. Distractible Difficult to console or comfort Each of the five categories (F) face; (L) legs; (A) Activity; (C) Cry; (C) Consolability is scored from 0-2, which results in a total score between 0 and 10.
* A child with a score of more than 4 on FLACC will receive intravenous acetaminophen 15mg/kg.
* The incision will then be monitored for signs of infection (Redness, Hotness, Swelling, Discharge, or Separation/Breakdown of deep tissues).
* Data regarding the incision will be obtained on day 7 postoperative or with sutures removal or any time before this if he/she develops any of wound inflammation signs earlier.

D) Measurements:

* Postoperative vital signs/hour for 4 hours.
* Faces Legs Activity Cry Consolability tool (FLACC, 0- 10) at 15 min, 1, and 3 h after operation.(11)
* Timing of first postoperative complaint of pain, first requirement for postoperative analgesia and total consumption of analgesia
* Laboratory measurements: white blood cells count at day 0 and day 7 postoperative.
* Culture: with first dressing change at day 7 postoperative from the wounds with discharge (suspected infected wounds).
* Wound infection and healing scale: using Southampton scoring system,(12) which classifies wounds according to healing into 6 grades (0, I, II, III, IV, V).

Table (II): Southampton wound scoring system Southampton wound scoring system Grade Appearance 0 Normal healing I Normal healing with bruising or mild erythema A Some bruising B Considerable bruising C Mild erythema II Erythema +other signs of inflammation A At one point B Around the sutures C Along the wound D Around the wound III Clear or heamoserous discharge A At one pint only (<2cm) B Along the wound (>2cm) C Large volume D Prolonged (3days) Major complication IV pus A At one point only (<2cm) B Along the wound (>2cm) V: deep or severe wound infection with or without tissue break down; hematoma requiring aspiration.

ETHICS OF RESEARCH

Research on human or human products:

Prospective study: Informed consent will be taken from patients. In case of incompetent patients the informed consent will be taken from the guardians.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 months-1 year
* Admitted for elective inguinal herniotomy surgery.

Exclusion Criteria:

* History of developmental delay or mental retardation.
* Diabetes mellitus type I.
* Known allergy or contraindication to any local anesthetics.
* Known congenital anomaly in the inguinal region.
* Any patient who will develop any infections postoperatively (respiratory infection, urinary infection) other than wound infection will be excluded.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Wound healing will be assessed and will be given grades 0-5 | 7 days
  Wound healing will be assessed and will be given grades 0-5

SECONDARY OUTCOMES:
Pain score (Faces) | one day.
  Faces 0-2
Pain score (Legs) | one day.
  Legs 0-2
Pain score (Activity) | one day.
  Activity 0-2
Pain score (Cry) | one day.
  Cry 0-2
Pain score (Consolability) | one day.
  Consolability 0-2

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hazem I Ahmad Sabry, MB,ChB MD, Principal Investigator — Alexandria Univeristy; Ramadan A Ammar, MB,ChB MD, Study Director — Alexandria Univeristy; Rana Bakr, MB,ChB, Principal Investigator — Alexandria Univeristy
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

REFERENCES:
- [Background] Eldor J. The antibacterial and antifungal effects of bupivacaine wound analgesia. JNYSORA 2009; 14:1-14.
- [Background] Johnson SM, Saint John BE, Dine AP. Local anesthetics as antimicrobial agents: a review. Surg Infect (Larchmt). 2008 Apr;9(2):205-13. doi: 10.1089/sur.2007.036. PMID 18426354
- [Background] Anaethesia UK. Pharmacology of regional anaesthesia. Anaethesia UK [Last Updated: 19 Nov, 2009]. Available from: http://www.frca.co.uk/article.aspx?articleid=100816. [Accessed on: 16 May, 2016].
- [Background] Silvani P, Camporesi A, Agostino MR, Salvo I. Caudal anesthesia in pediatrics: an update. Minerva Anestesiol. 2006 Jun;72(6):453-9. PMID 16682915
- [Background] Association of Paediatric Anaesthetists of Great Britain and Ireland. Good practice in postoperative and procedural pain management, 2nd edition. Paediatr Anaesth. 2012 Jul;22 Suppl 1:1-79. doi: 10.1111/j.1460-9592.2012.03838.x. No abstract available. PMID 22817132
- [Background] Fell D, Derrington MC, Taylor E, Wandless JG. Paediatric postoperative analgesia. A comparison between caudal block and wound infiltration of local anaesthetic. Anaesthesia. 1988 Feb;43(2):107-10. PMID 3354802
- [Background] Lao OB, Fitzgibbons RJ Jr, Cusick RA. Pediatric inguinal hernias, hydroceles, and undescended testicles. Surg Clin North Am. 2012 Jun;92(3):487-504, vii. doi: 10.1016/j.suc.2012.03.017. PMID 22595705
- [Background] Johr M. Regional anaesthesia in neonates, infants and children: an educational review. Eur J Anaesthesiol. 2015 May;32(5):289-97. doi: 10.1097/EJA.0000000000000239. PMID 25693139
- [Background] Polaner DM, Taenzer AH, Walker BJ, Bosenberg A, Krane EJ, Suresh S, Wolf C, Martin LD. Pediatric Regional Anesthesia Network (PRAN): a multi-institutional study of the use and incidence of complications of pediatric regional anesthesia. Anesth Analg. 2012 Dec;115(6):1353-64. doi: 10.1213/ANE.0b013e31825d9f4b. Epub 2012 Jun 13. PMID 22696610
- [Background] Cook TM, Counsell D, Wildsmith JA; Royal College of Anaesthetists Third National Audit Project. Major complications of central neuraxial block: report on the Third National Audit Project of the Royal College of Anaesthetists. Br J Anaesth. 2009 Feb;102(2):179-90. doi: 10.1093/bja/aen360. Epub 2009 Jan 12. PMID 19139027
- [Background] Crellin D, Sullivan TP, Babl FE, O'Sullivan R, Hutchinson A. Analysis of the validation of existing behavioral pain and distress scales for use in the procedural setting. Paediatr Anaesth. 2007 Aug;17(8):720-33. doi: 10.1111/j.1460-9592.2007.02218.x. PMID 17596217
- [Background] Bailey IS, Karran SE, Toyn K, Brough P, Ranaboldo C, Karran SJ. Community surveillance of complications after hernia surgery. BMJ. 1992 Feb 22;304(6825):469-71. doi: 10.1136/bmj.304.6825.469. PMID 1547415